CLINICAL TRIAL: NCT02110290
Title: Effects of Adapted Skiing and Snowboarding on Quality of Life in Children With Physical Disabilities
Brief Title: Effects of an Adapted Ski/Snowboarding Program on Quality of Life in Children With Physical Disabilities
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 10-1111
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Palsy; Traumatic Brain Injuries; Spinal Cord Injuries; Physical Disability
Keywords: quality of life; adaptive sports; therapeutic recreation; mental health
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries, Traumatic; Spinal Cord Injuries; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with Physical Disabilities: This group includes children 8-18 years old participating in an adapted ski/snowboarding program with any type of physical disability, including cerebral palsy, traumatic brain injury, spinal cord injury, and amputation.

SUMMARY:
This study is assessing quality of life in children with a physical disability who participate in the Children's Hospital Colorado Hospital Sports Program (HSP), where children with physical disabilities are able to participate in more organized sports and active programs with the use of adaptive equipment. This study would assess a child's self reported and parent perceived quality of life before and after child participation in HSP for the winter season. The investigators aim to determine the level of child and parent happiness and satisfaction in specific quality of life aspects including: physical activities and health, feelings, moods, self perception, home life, friends, school, learning and bullying. The investigators believe that children with any physical disability will have a more satisfactory reported quality of life after participating in HSP for one or many years.

DETAILED DESCRIPTION:
The purpose of this proposed research is to quantify the impact of participation in an adaptive ski/snowboarding program on parent perceived and child self-reported health related quality of life. To this effect, the study will assess children's self-perception of psychological, emotional, physical health of participants as well as their parents perception of the same, through the use of a validated self reported quality of life questionnaire, KIDSCREEN-52, before and after participating in an adaptive ski/snowboarding program every year.

Primary Aims:

1. To determine the level of subject and parent satisfaction and happiness, through a composite of 10 aspects in a quality of life questionnaire, following participation in the Children's Hospital Colorado Hospital Sports Program (HSP) for one winter season.
2. To determine the long-term impact of repeated participation in an adapted ski/snowboarding program through a composite of 10 aspects in a quality of life questionnaire, following participation in the Children's Hospital Colorado Hospital Sports Program (HSP) for consistent winter seasons.

ELIGIBILITY:
Inclusion Criteria:

* Physical disability
* Participant of HSP program

Exclusion Criteria:

* Completed parent and child KIDSCREEN questionnaires are not received before the subject's first day of skiing or snowboarding with the program
* Completed parent and child KIDSCREEN questionnaires are not received within 3 months after subject's completed participation with the program for that winter season

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Hospital Sports Program at Children's Hospital Colorado only has the capability to accommodate 60 to 65 children a year. This study contacts all of the subjects who meet the study inclusion criteria from the enrolled HSP participant list. It should be noted that the investigators will only be recruiting from children already participating in HSP; they will not be recruiting for children to join HSP.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2010-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Physical Wellbeing | Up to 5 years after study enrollment
  Short-term and long-term changes in the physical wellbeing assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
Psychological Wellbeing | Up to 5 years after study enrollment
  Short-term and long-term changes in the psychological wellbeing assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
Moods and Emotions | Up to 5 years after study enrollment
  Short-term and long-term changes in the moods and emotions assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
Self Perception | Up to 5 years after study enrollment
  Short-term and long-term changes in the self perception assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
Autonomy | Up to 5 years after study enrollment
  Short-term and long-term changes in the autonomy assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
Parents | Up to 5 years after study enrollment
  Short-term and long-term changes in the feelings towards parents assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
Financial | Up to 5 years after study enrollment
  Short-term and long-term changes in the feelings towards finance assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
Peers | Up to 5 years after study enrollment
  Short-term and long-term changes in the feelings towards peers assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
School | Up to 5 years after study enrollment
  Short-term and long-term changes in the feelings toward school assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.
Bullying | Up to 5 years after study enrollment
  Short-term and long-term changes in the feelings toward bullying assessed by both the child and parent in the questionnaire will be compared. The pre-season and post-season questionnaires from the same ski season will be used to compare changes after participation in one season. The earliest pre-season questionnaire and most recent post-season questionnaire will be compared to evaluate long-term changes.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Chang, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States